CLINICAL TRIAL: NCT05240118
Title: Risk Factors of Short-term and Long-term OUtcome in DIscharged Patients With Heart Failure With Mildly Reduced Ejection Fraction
Brief Title: Outcome of Discharged HFmrEF Patients
Acronym: OUDI-HF
Status: Completed | Type: Observational
Sponsor: Xiangtan Central Hospital (Other)
Responsible Party: Principal Investigator, Jianping Zeng, Dean, Xiangtan Central Hospital ,Director of cardiovascular clinic, Clinical Professor, Xiangtan Central Hospital
Other Study IDs: 2021/12
Record Dates: First submitted 2021-12-03; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure With Mid Range Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HFmrEF Group: HFmrEF (Heart failure with mildly reduced ejection fraction): ESC Guideline heart failure 2021: patients with LVEF 41-49%.
  non-cardiac events group versus cardiac events (cardiac death or heart failure-related rehospitalization) group

SUMMARY:
This study aimed to define the independent risk factors related cardiac events (cardiac death or heart failure-related hospitalization) among heart failure with mildly reduced ejection fraction (HFmrEF) patients who discharged from the Xiangtan Central Hospital. Through the long-term follow-up the cardiovascular outcome of patients being discharged from the hospital, the risk factors related to cardiovascular outcome (cardiac death or heart failure-related hospitalization) will be explored to provide clinical evidence to intervene the discharged HFmrEF patients aiming to improve patients outcome in the future clinical practice.

DETAILED DESCRIPTION:
This study aimed to define the independent risk factors related cardiac events (cardiac death or heart failure-related hospitalization) among heart failure with mildly reduced ejection fraction (HFmrEF) patients who hospitalized in Xiangtan Central Hospital from January 1, 2015 to August 31, 2020. The patients would be clinically followed-up until August 31, 2021 per clinical visit or telephone call, the risk factors related to cardiovascular outcome (cardiac death or heart failure-related hospitalization) will be explored to provide clinical evidence to intervene the discharged HFmrEF patients aiming to improve patients outcome in the future clinical practice.

The clinical features of hospitalized heart failure with mildly reduced ejection fraction (HFmrEF, EF 41-49%) will be analyzed by retrospectively by reviewing patients medical records, laboratory and clinical imaging examination results during initial hospitalization, clinical outcome of enrolled patients will be obtained through clinical visit and telephone call. The primary endpoint is the composite cardiac events (cardiac death or heart failure related rehospitalization). The secondary endpoint is the all-cause death.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Heart failure with mildly reduced ejection fraction (HFmrEF) Presence of symptoms and/or signs of HF, and a mildly reduced LVEF (41- 49%); Elevated natriuretic peptides (BNP >35 pg/mL or NT-proBNP >125 pg/mL); Other evidence of structural heart disease.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who attended the Xiangtan Cengtral Hospital in the time period between January 1, 2015 and August 31, 2020 with the diagnosis of HFmrEF.
Sampling Method: Non-Probability Sample
Enrollment: 1693 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Long-term risk factors related to cardiac events (cardiac death or heart failure-related rehospitalization) in discharged patients with heart failure with mildly reduced ejection fraction | The last patients would be clinically followed-up until August 31, 2021 per clinical visit or telephone call.
  Primary Outcome Measure:
  1.Long-term risk factors related to cardiac events (cardiac death or heart failure-related rehospitalization) in discharged patients with heart failure with mildly reduced ejection fraction The clinical features of hospitalized heart failure with mildly reduced ejection fraction (HFmrEF, EF 41-49%) will be analyzed retrospectively by reviewing their medical records, laboratory and clinical imaging examination results during initial hospitalization, clinical outcome up to the study end will be obtained through clinical visit and telephone call.

SECONDARY OUTCOMES:
Long-term risk factors related to all-cause death in discharged patients with heart failure with mildly reduced ejection fraction | The last patients would be clinically followed-up until August 31, 2021 per clinical visit or telephone call
  1. Long-term risk factors related to all-cause death in discharged patients with heart failure with mildly reduced ejection fraction The clinical features of hospitalized heart failure with mildly reduced ejection fraction (HFmrEF, EF 41-49%) will be analyzed retrospectively by reviewing their medical records, laboratory and clinical imaging examination results during initial hospitalization, all-cause death up to the study end will be obtained through clinical visit and telephone call.

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Zeng, M.D., Principal Investigator — Xiangtan Central Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Z, Zhu Y, Chen S, Wu M, Huang H, Peng K, Zhang L, Zhao W, Peng X, Li N, Zhang H, Zhou Y, Peng Y, Fan J, Zeng J. Sex differences in patients with heart failure and mildly reduced left ventricular ejection fraction. Sci Rep. 2023 Apr 26;13(1):6832. doi: 10.1038/s41598-023-33733-8. PMID 37100821